CLINICAL TRIAL: NCT04644523
Title: Prospective Validation of 5 Items in Nailfold Dermoscopy to Predict a Normal Capillaroscopy in Raynaud's Phenomenon
Brief Title: Dermoscopy in Primary Raynaud's Phenomenon
Acronym: VASCUL-R
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200701
Record Dates: First submitted 2020-10-21; First posted 2020-11-25 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Raynaud Phenomenon
Keywords: Dermoscopy; Nailfold capillaroscopy
MeSH Terms: conditions — Raynaud Disease | interventions — Dermoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dermoscopy — dermoscopy is currently used in daily practice in dermatology, for melanoma screening. Dermoscopy will be used in this study on peri-ungueal area.
  This is a non-invasive and painless exam.

SUMMARY:
Raynaud's phenomenon (RP) is very frequent in general population (up to 10%). Nailfold capillaroscopy (NFC) is recommended for patients presenting RP, to eliminate systemic disease such as systemic sclerosis. NFC is not easily available in clinical practice. Dermoscopy, used for pigmentary skin lesion screening, may help to detect giant loops, hemorrhages or other capillaries anomalies. However, no study has evaluated the performance of dermoscopy in primary RP. The objective is to determinate which items in dermoscopy are correlated with a normal NFC and predict with a good negative predictive value, a normal NFC in RP patients. The secondary objective is to assess inter-observer reproducibility of dermoscopy in patients with RP.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is very frequent in general population (up to 10%). Nailfold capillaroscopy (NFC) is recommended for patients presenting RP, to eliminate systemic disease such as systemic sclerosis. NFC is not easily available in clinical practice. Dermoscopy, used for pigmentary skin lesion screening, may help to detect giant loops, hemorrhages or other capillaries anomalies. However, no study evaluated the performance of dermoscopy in primary RP. A preliminary study (Tenon Hospital) showed an interest of dermoscopy in primary and secondary RP, with a negative predictive value of dermoscopy of 100% for capillaroscopy.

This is a prospective, multicentric French study comparing dermoscopy and capillaroscopy in patients attending dermatology or vascular medicine departments for the first evaluation of a RP.

The objective is to determinate which items in dermoscopy are correlated with a normal NFC and predict with a good negative predictive value, a normal NFC in RP patients. The secondary objective is to assess inter-observer reproducibility of dermoscopy in patients with RP.

The main hypothesis is that a normal dermocopy on five items is highly predictive of a normal NFC.

During a first consultation for RP, NFC will be realized with a clinical exam and a biological test (antinuclear antibodies), as official recommendations. Dermoscopy of peri-ungueal area will be realized by another investigator, if possible during the same consultation. Photographs of all fingers, except thumbs, will be made and will be reviewed by another investigator of another center. There will be no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* first consultation for bilateral Raynaud's phenomenon (RP)
* Bilateral Raynaud's phenomenon affecting at least one finger of each hand defined by a paroxysmal syncopal phase on exposure to cold,
* Affiliated to the French health care systeme

Exclusion Criteria:

* age < 18 years
* Presence of unilateral RP where the capillaroscopy is normal regardless of the cause

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Raynaud's phenomenon requiring capillaroscopy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Dermoscopic items | November 2022
  To determine wich dermoscopic items predict normal capillaroscopy in a first-time attending RP.

SECONDARY OUTCOMES:
Photography | November 2022
  Reproducibility of dermoscopy for the 5 items: all photographs of dermoscopy will be reviewed by another investigator from another center.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No